CLINICAL TRIAL: NCT03520816
Title: The Effect of Early Physiotherapy on Biochemical Parameters in Major Burn Patients: A Burn Center's Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Murat Ali ÇINAR,MSc,PT, Resarch Asistant, Hasan Kalyoncu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-12
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Burns; Physiotherapy; Exercises
Keywords: Fibronectin; Prealbumin; Physiotherapy; Major Burns; biochemical parameters
MeSH Terms: conditions — Burns; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Burn Physiotherapy Protocol Group (Experimental): Patients in the treatment group have been received to the physiotherapy programme from the first day of their stay in the hospital.
  Interventions: Other: Burn Physiotherapy Protocol
- Control Group (No Intervention): The control group consisted of patients who could not receive physiotherapy due to various reasons.

INTERVENTIONS:
Other: Burn Physiotherapy Protocol — It consisted of parameters such as early mobilisation and ambulatory training, chest physiotherapy, and both active and passive normal joint movement exercises.
  Arms: Burn Physiotherapy Protocol Group

SUMMARY:
Background: This study planned to investigate the effect of early physiotherapy on biochemical parameters in major burn patients.

Methods: Ten women (50%) and 10 men (50%) aged 21-47 years old were included in our study. Participants were divided into two groups: one group was the treatment group and the other was the control group. In the treatment group, patients were admitted to the physiotherapy programme from the first day they have been hospitalised, in addition to their routine treatment (medical, surgery, etc.), for 4 days per week. It consisted of parameters such as early mobilisation and ambulatory training, chest physiotherapy, and both active and passive normal joint movement exercises. The days of treatment were determined as Tuesday, Wednesday, Thursday and Friday. Patients could not be treated on a Monday because that was surgery day. The control group consisted of patients who could not receive physiotherapy due to various reasons. All patients included in the study were evaluated weekly for 6 weeks after admission to the hospital. Parameters such as demographic information, characteristics of burn injury, C-reactive protein, fibronectin, transferrin and prealbumin were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Major burn injury (according to ABA)
* Conscious patients

Exclusion Criteria:

* Inhalation injury
* Various chronic disorders
* Organ dysfunctions

Ages: 21 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Fibronectin | Changes in fibronectin at 6 weeks later
  Blood test
Prealbumin | Changes in prealbumin at 6 weeks later
  Blood test
C-reactive protein | Changes in C-reactive protein at 6 weeks later
  Blood test
Transferrin | Changes in transferrin at 6 weeks later
  Blood test

CONTACTS AND LOCATIONS:
Overall Officials: MURAT ALİ ÇINAR, Msc, Principal Investigator — Hasan Kalyoncu University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Lee KC, Joory K, Moiemen NS. History of burns: The past, present and the future. Burns Trauma. 2014 Oct 25;2(4):169-80. doi: 10.4103/2321-3868.143620. eCollection 2014. PMID 27574647
- [Result] Mandell SP, Gibran NS. Early Enteral Nutrition for Burn Injury. Adv Wound Care (New Rochelle). 2014 Jan 1;3(1):64-70. doi: 10.1089/wound.2012.0382. PMID 24761346
- [Result] Gillenwater J, Garner W. Acute Fluid Management of Large Burns: Pathophysiology, Monitoring, and Resuscitation. Clin Plast Surg. 2017 Jul;44(3):495-503. doi: 10.1016/j.cps.2017.02.008. Epub 2017 Apr 14. PMID 28576238
- [Result] Chinese Burn Association; Chinese Association of Burn Surgeons; Cen Y, Chai J, Chen H, Chen J, Guo G, Han C, Hu D, Huan J, Huang X, Jia C, Li-Tsang CW, Li J, Li Z, Liu Q, Liu Y, Luo G, Lv G, Niu X, Peng D, Peng Y, Qi H, Qi S, Sheng Z, Tang D, Wang Y, Wu J, Xia Z, Xie W, Yang H, Yi X, Yu L, Zhang G; Chinese Burn Care and Rehabilitation Association. Guidelines for burn rehabilitation in China. Burns Trauma. 2015 Oct 21;3:20. doi: 10.1186/s41038-015-0019-3. eCollection 2015. PMID 27574666
- [Result] Luzzani A, Polati E, Dorizzi R, Rungatscher A, Pavan R, Merlini A. Comparison of procalcitonin and C-reactive protein as markers of sepsis. Crit Care Med. 2003 Jun;31(6):1737-41. doi: 10.1097/01.CCM.0000063440.19188.ED. PMID 12794413